CLINICAL TRIAL: NCT00405691
Title: A Prospective, Multi-Center Clinical Study to Assess the Saftey and Effectiveness of the Impliant TOPS System
Brief Title: Safety and Effectiveness Study of the TOPS System, a Total Posterior Arthroplasty Implant Designed to Alleviate Pain Resulting From Moderate to Severe Lumbar Stenosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impliant, Ltd. (Industry)
Responsible Party: Dan Finan, Impliant, Inc.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TOPS-US-IDE-002
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-01

CONDITIONS: Low Back Pain; Leg Pain; Spondylolisthesis; Lumbar Spinal Stenosis
Keywords: Medical Device; Spine; Lumbar Spinal Stenosis; Degenerative Spondylolisthesis; Facet Arthrosis; Back and Leg Pain; Spine Research; Medical Device Research; Impliant; Lumbar Treatment; Spinal Treatment; Spinal Device
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: "TOPS System" - Total Posterior Arthroplasty Implant

SUMMARY:
The purpose of this multi-center, randomized, clinical study is to establish the safety and effectiveness of the TOPS™ System, used following decompression, in the treatment of lower back and leg pain with, or without spinal claudication, that results from moderate or severe lumbar spinal stenosis at one vertebral level between L3 and L5.

DETAILED DESCRIPTION:
This study is being conducted to evaluate a new surgical implant (TOPS™ System, Impliant). The TOPS™ System is an alternative to spinal fusion that is designed to stabilize but not fuse the affected vertebral level following decompression surgery to alleviate pain stemming from moderate/severe lumbar spinal stenosis while maintaining range of motion.

When non-surgical treatment is ineffective, decompression (including laminectomy and medial facetectomy) and fusion of the spinal segments with moderate/severe lumbar spinal stenosis has been used to stabilize the motion segment and to alleviate the patient's clinical symptoms. Spinal fusion surgery using metal instrumentation is designed to stop motion at a painful, unstable spinal segment by permanently fusing the segment. While fusion may decrease pain generated at the treated segment, the procedure also eliminate motion at the implanted level and transfers and thus increases loads on the adjacent segments.

The TOPS System is intended to provide stabilization following decompression in patients with disease at one level from L3 to L5. The ideal goal of stabilization is to preserve mobility but eliminate abnormal motion and prevent deformity. By using the TOPS System, it may be possible to preserve load-bearing dynamics and spinal biomechanics, and thereby maintaining motion at the treated segment.

The TOPS surgical technique, utilizing a standard top loading pedicle screw-based system, is the same as a standard posterior spinal fusion with the exception of the placement of the TOPS motion segment. Therefore, the surgeon will be executing the steps of surgical exposure, decompression, insertion of pedicle screws (with attention to proper placement/alignment) and closure in the same manner as he/she would in a standard posterior spinal fusion.

The objective of the clinical investigation is to compare the safety and effectiveness of the TOPS System to a control group of patients undergoing posterior spinal fusion with pedicle screws and local autograft bone in the treatment of back and leg pain that results from moderate/severe lumbar spinal stenosis at a single vertebral level between L3 to L5.

Prior to entering the study, patients will be evaluated by the investigator according to the inclusion/exclusion criteria. Patients recruited to the study will be randomized in a 1:1 ratio to undergo implantation of the TOPS System or the control spinal fusion procedure. Patient follow-up will be evaluated immediately post-operatively and at discharge, 6 weeks, 3 months, 6 months, 12 months, and 24 months.

ELIGIBILITY:
INCLUSION CRITERIA:

* Moderate to Severe lumbar spinal stenosis at a single level* between L3 - L5, with radiographic confirmation of any one of the following on CT, MRI, plain x-ray or myelography:

  * Evidence of thecal sac and/or cauda equina compression
  * Evidence of nerve root impingement by either osseous or non-osseous elements;
  * Evidence of hypertrophic facets with canal encroachment Moderate/severe spinal stenosis is further defined radiographically as;
  * moderate canal stenosis is a 25-49% reduction in the A/P dimension of the central and/or lateral foramen when compared to adjacent (cephlad) level
  * Severe canal stenosis is defined as 50% or greater reduction in the A/P dimension of the central and/or lateral foramen when compared to the adjacent (cephlad) level **Patients which require minimal decompressive surgery at an adjacent level, may have a laminonotmy or soft tissue resection as long as the decompression does not compromise the stability of the adjacent segment.
* At least six (6) months of failed, conservative treatment prior to surgery, including physical therapy, use of anti-inflammatory medications at maximum specified dosage; administration of epidural/facet injections.
* Age 40-75 years old (male or female).
* Up to one prior surgery without instrumentation implanted at any lumbar vertebral level limited to the following:

  * IDET,
  * laminotomy,
  * laminectomy,
  * foraminotomy
  * Discectomy (that occurred at least three years ago without any reoccurrence of herniation)
* Lower back pain and/or sciatica with or without spinal claudication.
* VAS leg pain of at least 40/100 at baseline.
* Oswestry Questionnaire score of at least 40/100 at baseline.

EXCLUSION CRITERIA:

* Back or non-radicular leg pain of unknown etiology
* Spondylolisthesis Grade II or higher
* Stenosis caused by an extruded spinal disc fragment
* Lytic spondylolisthesis
* More than one (1) motion segment involved in the degenerative pathology to the extent that justifies its inclusion in the surgical procedure, unless a decompression alone can be done at that level without compromising stability.
* Known allergy to titanium and/or polyurethane
* Prior fusion surgery at any lumbar vertebral level with or without instrumentation
* Supplemental interbody support required (e.g., bone graft, spacers, VBRs, or fusion cages)
* Clinically compromised vertebral bodies at the affected level(s) due to any traumatic, neoplastic, metabolic or infectious pathology.
* Scoliosis of greater than ten (10) degrees (both angular and rotational)
* Morbid obesity defined as a body mass index > 40 or a weight more than 100 lbs. over ideal body weight.

Note: Additional inclusion/exclusion criteria are applied. Please contact Impliant for further details.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2006-09

PRIMARY OUTCOMES:
Primary safety and effectiveness to determine patient success are: 1 .15% ODI improvement vs baseline at 24 mos; 20 mm leg and back pain VAS improvement vs baseline at 24 mos.
2. improvement of at least 20 mm in leg pain at 24 months compared to baseline using a VAS pain scale;
3. maintenance or improvement of neurological status;
4. no revisions, supplemental fixation, and removals;
5. absence of major device-related complications (device component degradation or breakage, device component separation or disassembly, device component loosening (including screw loosening)) requiring revisions, supplemental fixation, and removals;
6. absence of spontaneous fusion in the investigational group and lack of fusion in the control

SECONDARY OUTCOMES:
Secondary outcome measurements that will be assessed include: 1. Zurich Claudication Questionaire scores, SF-36 scores, and VAS back pain score
2. Adverse events
3. time to recovery, work status, OR time, blood loss, and pharmaceutical use
4. radiographic measurements (degree of stenosis & spondylolisthesis, disc height, disc angle, alignment, translational motions, Range of Motion (affected level and entire lumbar spine), disc health (affected & adjacent levels), fusion status.

CONTACTS AND LOCATIONS:
Overall Officials: Paul McAfee, M.D., Principal Investigator — Orthopaedic Associates, P.A
Locations (16):
- United States (16):
  - Institute for Advanced Spinal Research In California, Beverly Hills, California
  - Century City Doctors Hospital, Beverly Hills, California
  - Seton Medical Center, Daly City, California
  - Yale University - School of Medicine, New Haven, Connecticut
  - The Orthopaedic & Sports Medicine Ctr., Trumbull, Connecticut
  - Florida Orthopaedic Institute, Tampa, Florida
  - Illinois Neuro Spine Center, Ogden, Illinois
  - Saint Joseph Medical Center & Orthopaedic Associates, Baltimore, Maryland
  - The Boston Spine Group, Boston, Massachusetts
  - New England Neuro Assoc., Springfiled, Massachusetts
  - Columbia Orthopedic Group, Columbia, Missouri
  - Orthopedic Spine Care of Long Island, Huntington Station, New York
  - Buffalo Spine Surgery, Lockport, New York
  - Carolinas Medical Center Hospital - Neurosurgery & Spine Associates, Charlotte, North Carolina
  - NeuroSpine Center of Wisconsin, Appleton, Wisconsin
  - Milwaukee Spinal Specialists, Milwaukee, Wisconsin